CLINICAL TRIAL: NCT05494918
Title: A Phase I, Multi-center, Open-label, Dose Escalation, First-In-Human Study to Assess the Safety, Tolerability and Pharmacokinetics of JSKN003 in Subjects With Advanced or Metastatic Solid Malignant Tumors
Brief Title: First-In-Human Study in Subjects With Advanced or Metastatic Solid Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alphamab (Australia) Co Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JSKN003-101
Record Dates: First submitted 2022-08-04; First posted 2022-08-10 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors; Metastatic Solid Tumors

STUDY DESIGN:
Intervention Model Description: The starting dose of JSKN003 is 1.0 mg/kg, followed by 2.1, 4.2, 5.3, 6.3, 7.3, 8.4, 9.4 and 10.5 mg/kg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose escalation (Experimental): It's a dose escalation to identify the Maximum Tolerated dose (MTD) , recommended dose for expansion (RDE) or recommended Phase II dose (RP2D) of JSKN003, guided by the modified ADT design and BOIN design.
  Interventions: Drug: JSKN003

INTERVENTIONS:
Drug: JSKN003 — JSKN003 is to be administered via intravenous (IV) dose
  Other Names: anti-Her2 ADC JSKN003

SUMMARY:
This study is an open-label, multicenter, first-in-human, Phase I, dose escalation study to evaluate the safety, tolerability, PK, and preliminary anti-tumor activity of JSKN003 in subjects with advanced inoperable or metastatic solid malignant tumors that are expected to be HER2 expression.

DETAILED DESCRIPTION:
The dose escalation study will utilize single patient accelerated dose titration for the first two dose levels, 1.0 and 2.1 mg/kg, followed by dose cohorts 4.2, 5.2, 6.3, 7.3, and 8.4 mg/kg which will all be enrolled and monitored using the Bayesian optimal interval design, aimed at determining the MTD, RDE/RP2D of JSKN003. The dose-escalation of 9.4 mg/kg and 10.5 mg/kg should be determined per discussion between Safety Monitoring Committee and sponsor if deemed necessary, the SMC had the right of deciding to dose-escalate at other dose levels . Moreover, the SMC is also responsible for deciding the MTD and the recommended dose level for dose-expansion study.

Enrolled patients will be sequentially assigned to the planned dose levels as required by the protocol and treated with JSKN003 IV Q3W to observe the occurrence of treatment related AEs and dose limiting toxicities. The DLT observation period is 21 days from administration of the first dose of JSKN003.

The study will use a modified ADT design and BOIN design for dosing cohort management to determine the MTD and RDE/RP2D. The starting dose of JSKN003 is 1.0 mg/kg, followed by 2.1, 4.2, 5.3, 6.3, 7.3, 8.4, 9.4 and 10.5 mg/kg. The investigational product will be administered on Day 1 every 3 weeks via intravenous infusion, and the first cycle of JSKN003 treatment is for DLT evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide signed informed consent form (ICF) for the trial.
2. Male or female, 18 years of age or older; willing and able to comply with study requirements.
3. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1 with no deterioration within 2 weeks of scheduled study treatment, and life expectancy ≥ 12 weeks.
4. Must have a pathologically documented advanced/unresectable or metastatic solid malignant tumor with HER-2 expression (IHC ≥ 1+) that is refractory to or intolerable with standard treatment, or for which no standard treatment is available.
5. Baseline measurable disease according to RECIST 1.1. Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Adequate organ function assessed within 7 days prior to first trial treatment [had not received blood transfusion, erythropoietin (EPO), granulocyte colony stimulating factor (G-CSF) or other relevant medical support within 14 days before the administration of the investigational product].
7. Have adequate treatment washout period before first trial treatment.
8. Have LVEF ≥ 50% by either echo cardiography (ECHO) or multiple-gated acquisition (MUGA) within 28 days prior to first trial treatment.
9. Female or male subjects of childbearing potential should be willing to use a highly effective method of contraception (with a failure rate of less than 1.0% per year) from first study treatment to 180 days after completion of the trial treatment. Female of childbearing potential should have a negative pregnancy test within 7 days prior to first trial treatment (childbearing potential is defined as premenopausal females without documented tubal ligation or hysterectomy, or postmenopausal females within 1 year).

Exclusion Criteria:

1. Clinically active central nervous system (CNS) metastases, defined as untreated and symptomatic, with following exceptions:

   * Clinically stable through MRI/CT scans (at least 2 consecutive scans within prior 6 months including 1 scan within 28 days prior to screening) and no progressive or uncontrolled neurologic symptoms or signs (e.g., seizures, headaches, central nausea/emesis, progressive neurologic deficits, papilledema) for at least 4 weeks prior to the first treatment.
   * Any untreated asymptomatic brain metastases not requiring immediate local or systemic therapy (e.g., mannitol or corticosteroids).
   * Leptomeningeal metastasis is excluded from the study entry.
2. Concurrent malignancy within 5 years prior to entry other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma, prostate cancer, thyroid cancer not requiring treatment, ductal carcinoma in situ of the breast, or <T1 urothelial carcinoma.
3. Prior treatment with an antibody-drug conjugate (ADC) which consists of a topoisomerase I inhibitor derivative.
4. History of uncontrolled intercurrent illness including but not limited to:

   * Active HBV or HCV infection. If HBsAg and HCV antibody positive, HBV DNA and HCV RNA assay should be performed. Subjects are eligible if HBV DNA ≤ 500 UI/ml (or 2000 copies/ml) or HCV RNA negative.
   * Known HIV infection or known history of acquired immune deficiency syndrome (AIDS);
   * Active tuberculosis infection.
   * Active infection within 4 weeks prior to the first dose of trial treatment that require the use of systemic antibiotics ≥ 7 days.
   * Hypertension uncontrolled by standard therapies (not stabilized to 160/100 mmHg);
   * Clinically significant (that is, active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina pectoris (< 6 months prior to enrolment), congestive heart failure (New York Heart Association Classification Class II-IV) or serious cardiac arrhythmia requiring medication (including corrected QT interval prolongation of > 470 msec for women and > 450 for men calculated according to Fridericia and/or pacemaker or prior diagnosis of congenital long QT syndrome;
   * Serious nonhealing wound, ulcer or bone fracture.
5. Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids or current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by image at screening.
6. Previous severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) infection either suspected or confirmed within 4 weeks prior to screening. Acute symptoms will be excluded, or must have resolved and based on investigator assessment, there are no sequela that would place participant at a higher risk of receiving investigational treatment.
7. Subjects with ascites, pleural effusion, pericardial effusion which cannot be controlled by appropriate interventions.
8. Have unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia, grade 2 hypoparathyroidism) related to prior anticancer therapy and stable anemia (i.e., untransfused Hb ≥ 9 g/dL without the need for supportive transfusion within 2 weeks of screening) not yet resolved to grade ≤ 1 (NCI-CTCAEV5.0).
9. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses ≤ 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. A brief course of corticosteroids for the prophylaxis (e.g., contrast dye allergy) or treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
10. History of life-threatening hypersensitivity or known to be allergic to protein drugs or recombinant proteins or excipients in JSKN003 drug formulation.
11. Prior history of Herceptin induced anaphylaxis, angioedema, or severe hypotension.
12. Other conditions that, in the investigators' opinion, would make subjects inappropriate to participate in this study, such as a history of mental illness, alcoholism or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
MTD | Postdose of last participant up to 1 year
  Maximum tolerated dose
Preliminary RDE/RP2D | Postdose of last participant up to 1 year
  recommended dose for expansion / recommended phase 2 dose
DLTs | Baseline up to 21 days after the first dose
  Dose Limiting Toxicities
Adverse Events | Baseline up to 30 days after the last dose of study drug, up to 1 year
  Incidence and severity of treatment-emergent adverse events (TEAEs), treatment-related adverse events (TRAEs), serious adverse events (SAEs)

SECONDARY OUTCOMES:
Cmax of JSKN003 | Post last dose up to Day 90
  Maximum (Peak) Observed blood Concentration (Cmax) of JSKN003 Following First Dose
Tmax of JSKN003 | Post last dose up to Day 90
  Time of Maximum blood Concentration (Tmax) of JSKN003 Following First Dose
AUC of JSKN003 | Post last dose up to Day 90
  The blood PK parameters of JSKN003 and its analytes for area under the concentration-versus-time curve from time 0 to the last quantifiable concentration as calculated by the linear-up log-down trapezoidal method (AUClast) and AUC from time 0 to infinity (AUCinf) elimination rate constant associated with the terminal phase were estimated using standard non-compartmental methods.
Terminal Elimination Half-life (t1/2) | Post last dose up to Day 90
  The blood PK parameters of Terminal elimination half-life for JSKN003
ORR | Postdose of last participant up to 1 year
  Objective response rate (ORR) by independent central review was defined as the proportion of participants who achieve either complete response [CR] or partial response [PR] per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
TTR | Postdose of last participant up to 1 year
  TTR is defined as the time from the date of first study dose to the date of earliest qualifying response
DoR | Postdose of last participant up to 1 year
  Duration of response for responders (CR or PR) is defined as the time interval between the date of earliest qualifying response and the date of PD or death for any cause, whichever occurs earlier.
PFS | Postdose of last participant up to 1 year
  PFS is defined as the time from the date of first study dose to disease progression or death whichever occurs first. Subjects without event (no disease progression or alive at last visit) will be censored at the date of "last tumor assessment".
Anti-JSKN003 antibody | Post last dose up to Day 90
  Status (positive or negative) and serum titers of anti-JSKN003 antibody

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Chan, Principal Investigator — Breast Cancer Research Centre-WA,Hollywood Consulting Centre
Locations (1):
- Breast Cancer Research Centre, Perth, Western Australia, Australia